CLINICAL TRIAL: NCT00508534
Title: An Open-Label Study to Evaluate the Effects of Repeat Dosing of Esomeprazole on the Pharmacokinetics of SB-751689 in Healthy Adult Subjects
Brief Title: A Study To Evaluate The Effects Of Repeat Dosing Of Esomeprazole On The Pharmacokinetics Of SB-751689 In Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR9106339
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Osteoporosis
Keywords: pharmacokinetic study,; gastric pH
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: SB-751689

SUMMARY:
This study will examine the effects of altering gastric pH in healthy volunteers on the pharmacokinetics of SB-751689 with or without food.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females between the ages of 21 and 55, inclusive, will be eligible for the study. Female subjects must be of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or bilateral oophorectomy or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/ml or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* The subject has a body mass index (BMI) of 19 to 31 kg/m2 where BMI= (weight in kg)/(height in meters)2
* Subjects must be genotyped as poor metabolizers or heterozygous extensive metabolizers for CYP2C19.
* The subject is capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Genotyped homozygous extensive metabolizers for CYP2C19 (Section 6.1.1 CYP2C19 Polymorphism Genotyping).
* Any clinically relevant abnormality identified on the screening history and physical or laboratory examination, 12-lead electrocardiogram (ECG) and/or 24 hour Holter, including QTc > or = 450 msec.
* Positive urine drug screen at screening.
* Positive urine test for alcohol at pre-dose.
* Positive for HIV at screening
* Chronic hepatitis B and C, as evidenced by positive Hepatitis B surface antigen or Hepatitis C antibody.
* Urinary cotinine levels indicative of smoking at screening.
* History of smoking or use of nicotine containing products within one year of the study or >10 pack-year history of smoking overall.
* History of regular alcohol consumption exceeding 7 units/week for women and 14 units/week for men (1 unit = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening.
* History of drug abuse within 6 months of the study.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity with 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of the current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or nonprescription drugs including antacids, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days or (14 days if the drug is a potential enzyme inducer or 5 half-lives, whichever is longer) prior to the first dose of study medication, unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study procedures or compromise subject safety.
* Consumption of red wine, grapefruit, grapefruit juice or grapefruit-containing products within 14 days prior to the first dose of study medication.
* Donation of blood in excess of 500 mL within 56 days prior to dosing.
* Evidence of renal, hepatic or biliary impairment
* History of serious gastrointestinal disease
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* History of clinically significant cardiovascular disease.
* History of pernicious anemia, pancreatitis, osteosarcoma or kidney stones.
* Medical conditions which might alter bone metabolism.
* Liver function tests (ALT, AST, GGT, alkaline phosphatase, total bilirubin) and/or parathyroid hormone (PTH) test or CPK outside the reference range at screening.
* Males unwilling to refrain from fathering a child during the study and for 14 days following the last dose of study medication.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2007-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Cmax and AUC of SB-751689 alone or after treatment with esomeprazole, and under fasted or fed conditions | over 1 week

SECONDARY OUTCOMES:
Adverse event report, ECGs, vital signs, laboratory test, and clinical monitoring | over a week

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Singapore, Singapore